CLINICAL TRIAL: NCT04653285
Title: Facilitating Motor Skill Learning by Aerobic Training in Parkinson's Disease III
Brief Title: Facilitating Motor Skill Learning in Parkinson's Disease III
Acronym: FaST-PD-III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: German Foundation for Neurology (Other); Klinik für Neurologie, Klinikum Würzburg Mitte, Standort Juliusspital (Unknown)
Responsible Party: Principal Investigator, Simon Steib, PhD, Principal Investigator, University of Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSN-2020
Record Dates: First submitted 2020-10-12; First posted 2020-12-04 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; motor learning; neuroplasticity; aerobic exercise; cardiovascular exercise; balance; postural instability; motor memory; consolidation
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- motor skill practice + aerobic exercise (Experimental): bout of aerobic exercise following motor skill practice
  Interventions: Behavioral: motor skill practice; Behavioral: aerobic exercise
- motor skill practice + rest (Active Comparator): seated rest following motor skill practice
  Interventions: Behavioral: motor skill practice; Behavioral: rest

INTERVENTIONS:
Behavioral: motor skill practice — Motor learning task on a stability platform (stabilometer). Participants try to keep the tiltable platform in a horizontal position in trials of 30s.
Behavioral: aerobic exercise — A bout of moderate intensity aerobic exercise on a cycle ergometer following motor skill practice.
  Arms: motor skill practice + aerobic exercise
Behavioral: rest — Seated rest following motor skill practice.
  Arms: motor skill practice + rest

SUMMARY:
The study is designed to assess the effects of cardiovascular (aerobic) exercise on motor skill learning in Parkinson patients. Specifically, the investigators examine whether moderate-intense aerobic exercise, performed immediately following motor skill practice over the course of a six week intervention period, facilitates motor memory consolidation. In this experimental trial, participants will be randomly allocated to either an intervention group (motor skill practice + aerobic exercise) or control group (motor skill practice + seated rest).

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurodegenerative disorder that is characterized by motor control impairments, such as gait disturbances and postural instability. Beneficial effects of exercise are attributed to mechanisms of neuroplasticity, and task-specific motor training (repeated practice of a skill) is consequently considered to be a motor learning process. Importantly, the formation (acquisition) and consolidation of motor memories is impaired in PD compared to healthy individuals of similar age.

Thus, it is crucial to identify strategies to enhance motor learning in people with PD. Recent studies have accumulated evidence to show that acute (single bouts of) and chronic (multiple bouts of) cardiovascular exercise can facilitate motor skill learning. However, this evidence is mainly derived from studying healthy individuals. In a first study including PD patients, the investigators recently found improved motor memory consolidation, but not improved skill acquisition, when practice was preceded by a single bout of cardiovascular exercise.

These results suggested that acute exercise may enhance motor memory formation processes, but could potentially interfere with motor skill acquisition when performed prior to practice. Consequently, in a second study the investigators examined whether performing a single bout of cardiovascular exercise immediately following skill practice would enhance motor memory consolidation without affecting skill acquisition in PD. The results of this second study suggested that even a single moderate intense bout performed immediately following skill practice improves motor memory consolidation in PD patients.

Going onward from the previous two studies, the present study will investigate the effects of performing cardiovascular exercise immediately following skill practice over the course of a six week intervention period on motor memory consolidation. It will be examined how the regular direct coupling of motor learning skill practice and cardiovascular exercise influences the consolidation and automation of the practiced movements.

In an experimental trial, participants will be randomly allocated to one of two groups. Both groups will practice balancing on a stability platform (motor learning task). The experimental group will additionally perform a bout of aerobic exercise (cycle ergometer) immediately following motor practice, while the control group will rest. This intervention will be held over a period of six weeks. Subsequently, motor skill retention will be tested seven days after the last training session.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease stage 1-3,5 on Hoehn & Yahr scale
* Ability to stand unaided and walk without an assistive device
* Stable medication during the study period
* Unfamiliar to the motor task (stabilometer)

Exclusion Criteria:

* On-off and wearing-off phenomena
* Unstable medical or psychiatric illness
* Clinically relevant cardiovascular or orthopaedic disease
* Severe polyneuropathy
* Cognitive impairment
* Smoking > 10 cigarettes/day
* Caffeine > 6 cups of coffee/day
* Alcohol > 50 g (two glasses)/day

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Time in balance | Week 1: performance at Baseline, Week 2 - 7: performance at practice session, Week 8: seven day retention performance
  Motor memory consolidation: Change of time in balance (angular displacement ±5° from horizontal) over the course of all six skill practice sessions and the seven day retention test.

SECONDARY OUTCOMES:
Root mean square error (RMSE) | Week 1: performance at Baseline, Week 2 - 7: performance at practice session, Week 8: seven day retention performance
  Memory consolidation: Change of root mean square error (average angular deviation from horizontal) over the course of all six skill practice sessions and the seven day retention test.
Dual-Task-Performance: Counting Backwards | Week 1: performance at baseline; Week 8: performance at seven day retention
  Motor memory automatization: Change of time in balance (angular displacement ±5° from horizontal) in addition to error score of a backwards-counting-task from Pre- to Post-Assessment
Transfer Test Performance: Fullerton Advanced Balance Scale (FAB - Scale) | Week 1: performance at baseline; Week 8: performance at seven day retention
  Transfer Effects of Balance: Change of the achieved score on the FAB - Scale from Pre- to Post- Assessment; minimum value: 0; maximum value: 40; higher scores indicate better outcome
Muscular Endurance: Five Times Sit to Stand Test | Week 1: performance at baseline; Week 8: performance at seven day retention
  Strength Endurance: Change of time necessary to rise five times from a chair
BDNF - Levels (Brain-derived neurotrophic factor) | Week 1: BDNF concentration at baseline; Week 2 a + b: BDNF concentration before (a) and after (b) Intervention; Session: 7 a + b: BDNF concentration before (a) and after (b) Intervention; Week 8: BDNF concentration at seven day retention
  Change of BDNF - Concentration in Blood samples
VO2 max Level | Week 1: VO2max at baseline; Week 8: VO2max at seven day retention
  Maximum oxygen uptake and overall effect on cardiovascular fitness level: submaximal stress test on bicycle ergometer
Unified Parkinson's Disease Rating Scale (UPDRS) - Motor Score | Week 1: score at baseline; Week 8: score at seven day retention
  Parkinson Disease Rating Score (motor section): Change of UPDRS Score; minimum value: 0; maximum value: 132; higher scores indicate worse outcome
Montreal Cognitive Assessment Score (MoCA - Score) | Week 1: score at baseline; Week 8: score at seven day retention
  Cognitive capability: Montreal Cognitive Assessment Score; minimum value: 0; maximum value: 30; higher scores indicate better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Simon Steib, Dr., Principal Investigator — Institute of Sport and Sport Science, Heidelberg University
Locations (1):
- Heidelberg University, Institute of Sport and Sport Science, Im Neuenheimer Feld 720, Heidelberg, Bade-Wuerttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: project website — https://www.sport.fau.eu/das-institut/forschung/bewegung-und-gesundheit/forschungsprojekte/optimierung-motorischer-lernprozesse-in-der-rehabilitation-von-parkinsonpatienten/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT04653285/Prot_SAP_000.pdf